CLINICAL TRIAL: NCT05724719
Title: Multimodal Prediction of Seizure Recurrence After Unprovoked First Seizure to Guide Clinical Decision-making: a Multi-centre Study of Cognition, Mood and Brain Connectivity As Predictors
Brief Title: Seizure Recurrence After Unprovoked First Seizure
Status: Recruiting | Type: Observational
Sponsor: Dr. Gavin Winston (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Dr. Gavin Winston, Dr. Gavin Winston, Associate Professor, Dept. of Medicine, Queen's University, Faculty-Centre for Neuroscience, Queens University, Queen's University
Organization: Queen's University (Other)
Other Study IDs: DMED-2681-22; PJT-183906 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Single Seizure; Epilepsy
Keywords: Cognition; Mood; Brain Connectivity; Neuroimaging; Neurophysiology
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Unprovoked First Seizure (UFS): Participants will undergo cognitive screening assessment, MRI imaging and EEG (if not already done) within 2-4 weeks of the initial First seizure clinic visit. Seizure recurrence will be monitored by a diary provided to each participant with details of the research team to contact in the event of a seizure. A researcher via perform telephone reminders at 3, 6, 9 and 12 months following the seizure. The primary outcome will be seizure recurrence at 12 months.
- Healthy Controls: Healthy control participants will complete the same neuropsychological battery, MRI scans and EEG protocols to evaluate baseline level of impairment in a healthy population and for the group comparisons of UFS to healthy controls to establish the changes already present at initial presentation with UFS.

SUMMARY:
One in 10 people have a seizure during their life. Usually no cause is identified. Seizures without an identified cause are called unprovoked first seizure (UFS). Most people with UFS do not have further seizures. Being able to predict the risk of more seizures as soon as possible would help doctors decide whether to suggest treatment after UFS.

Studies show that seizures are associated with changes in brain structure and function that are difficult to detect with standard assessments but can be detected with advanced techniques. Changes in connections between brain regions are also linked to subtle problems in thinking and mood.

The investigators will examine brain connections using detailed brain scans, thinking, and mood in people with UFS and develop an accurate method for calculating the risk of further seizures.

200 adult patients and 75 matched healthy controls from the Halifax and Kingston First Seizure Clinics will undergo cognitive screening assessment of major cognitive domains, MRI imaging including structural scans, resting-state functional MRI (rsfMRI) and diffusion-weighted imaging (DWI), and EEG.

Seizure recurrence will be assessed prospectively and a multimodal machine learning model will be trained to predict seizure recurrence at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* This study will consider adult patients between the ages of 18-65 years seen in the First Seizure Clinics in Halifax and Kingston with unprovoked first seizure.
* The investigators will also include a sample of age, sex, and education-matched healthy controls with the same exclusion criteria.

Exclusion Criteria:

* Individuals over the age of 65 will not be included to reduce the probability of including individuals with early dementia.
* The investigators will also exclude individuals who, upon assessment during their first clinic appointment, are determined to have non-epileptic events, recurrent events or diagnosis of epilepsy (e.g. based on abnormal CT or EEG), provoked seizure (e.g. medication, substance misuse, metabolic), acute symptomatic seizures, those with an existing prescription for antiseizure drugs, significant CNS comorbidity that may affect cognition and brain networks (e.g. progressive neurological disorder, MS), previous neurosurgery, or contraindication to MRI.
* Finally, although there is no known risk to a fetus from MRI scanning, as is standard in research studies involving MRI, pregnant participants will be excluded and those that suspect that they may be pregnant require a negative pregnancy test before scanning.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 years old with unprovoked first seizure; age, sex and education-matched healthy controls.
  Multi-centre, the study population will consist of adults from across Atlantic Canada, and South-Eastern Ontario.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Seizure Recurrence after Unprovoked First Seizure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gavin P Winston, BM BCh, PhD, Principal Investigator — Queen's University; Antonina Omisade, BA, PhD, Principal Investigator — Nova Scotia Health Authority
Locations (2):
- Canada (2):
  - Dalhousie University and Nova Scotia Health Authority, Halifax, Nova Scotia
  - Queen's University and Kingston Health Sciences Centre, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beattie BC, Batista Garcia-Ramo K, Biggs K, Boisse Lomax L, Brien DC, Gallivan JP, Ikeda K, Schmidt M, Shukla G, Whatley B, Woodroffe S, Omisade A, Winston GP. Literature review and protocol for a prospective multicentre cohort study on multimodal prediction of seizure recurrence after unprovoked first seizure. BMJ Open. 2024 Apr 5;14(4):e086153. doi: 10.1136/bmjopen-2024-086153. PMID 38582538